CLINICAL TRIAL: NCT00856479
Title: A Randomized Controlled Cost Study of Infuse BMP 2 vs Iliac Crest Autograft for Non Union of Long Bone Fractures
Acronym: Infuse
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study never started
Sponsor: Ross Leighton (Other)
Collaborators: Canadian Orthopaedic Trauma Society (Other)
Responsible Party: Sponsor-Investigator, Ross Leighton, Orthopedic Surgeon, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Infuse Study; COTS Grant
Record Dates: First submitted 2009-02-26; First posted 2009-03-05 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Non Union Diaphyseal Fractures
Keywords: Infuse; cost analysis; Non union diaphyseal fracture; The efficacy of Infuse BMP 2 in Non union diaphyseal fractures. Also the cost analysis with the amount of time spent in hospital post op.

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Infuse (Active Comparator): The patient will receive BMP 2 with allograft
  Interventions: Device: Infuse Bone Morphogenic Protein (BMP) 2
- 2 Iliac crest autograft (Active Comparator): Autograft from Patients Iliac Crest and allograft
  Interventions: Procedure: iliac crest autograft

INTERVENTIONS:
Device: Infuse Bone Morphogenic Protein (BMP) 2 — "Infuse" is a synthetic bone morphogenic protein which means it has the ability to help your bone to form and heal if inserted in the fracture site. "Infuse" may be the first commercially available product approved by Health Canada to accelerate the healing of long bone non-unions requiring surgical intervention.
  Arms: 1 Infuse
Procedure: iliac crest autograft — A piece of the patients iliac crest bone is take and mixed with bone from a bone bank to supplement the bone loss in the fracture
  Arms: 2 Iliac crest autograft

SUMMARY:
We are inviting individuals such as yourself, who have diaphyseal fracture (broken bone) with a non union to participate in this research study. A non-union is a lack of bone healing (bone growth where the break in the bone occurred) after 3 months after the operation. The diaphyseal is an area of a specific bone (usually near the middle) where the fracture occurred. The bones we are interested in are the clavicle (collar bone), tibia (lower leg), femur (upper leg), humerus (upper arm) and forearm (lower arm). Treatment goals for these types of fractures are to minimize later surgeries, to assist the healing process, and to decrease the time to healing. The ability of a patient with non-union (lack of bone healing after 3 months post operation) to return to the work force and to normal activities more quickly not only has a good financial impact on society (community), but also improves over-all physical and mental well-being of the patients.

"Infuse" is a synthetic bone morphogenic protein which means it has the ability to help your bone to form and heal if inserted in the fracture site. "Infuse" may be the first commercially available product approved by Health Canada to accelerate the healing of long bone non-unions requiring surgical intervention.

Although the safety and efficacy of Infuse has been demonstrated through numerous pre-clinical studies, further human clinical trial is needed to evaluate the safety and the power to produce effects of this product particularly with respect to non unions of long bones. The purpose of this study is to evaluate the safety and the power to produce effects of Infuse implanted during treatment of long bone non unions to reduce later surgeries required to augment the healing process and to accelerate the time to healing.

Given this, the orthopaedic community has planned this study in order to scientifically establish the most effective treatment method to restore function after this type of injury.

DETAILED DESCRIPTION:
We propose a multi-centre Canadian randomized Study wherein 80 patients are randomized (put in groups by no standard pattern ie. flipping a coin) to receive both autograft (sample of your own bone: iliac crest) and allograft (bone chips from bone bank) or "infuse" (synthetic bone morphogenic protein) and allograft using locked plates. Locked plates are surgical plates placed on the fracture in which the screws lock into the plate when they have been completely screwed into the bone through holes on the plate. Our objective is to assess the total cost of the patients treated in both study group and the benefits of the Infuse by comparing the new bone formation in the fracture site.

We will monitor critical aspects of operative care and rehabilitation at regular intervals, up to 2 year after surgery. We will independently monitor revision surgery (surgeries to repair a previous surgery) rates. We will also assess patients for functional health and quality of life outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for entry into the study:

a) Patients must require open surgical treatment of non-union of a diaphyseal fracture of the tibia, humerus, femur, radius or ulna sustained secondary to trauma.

c) Patients must be candidates for surgical treatment with an intramedullary nail or locked or unlocked plate.

d) Patients must have a fracture of the diaphysis as defined for that specific bone.

e) Patients must show radiographic evidence of skeletal maturity (closed epiphyseal plates).

Exclusion Criteria:

Patients with any of the following criteria, are not eligible for entry into the study:

1. Patients requiring mechanical fixation other than Intramedullary nailing or plating (i.e. no external fixation)
2. Patients with fractures that fall outside the diaphysis defined for the specific bone in question, i.e. no metaphyseal fractures.
3. Patients with segmental circumferential bone loss >4cm.
4. Patients whose fractures are the result of a tumour
5. Infection per se, does not result in exclusion but it must be treated and the soft tissue envelope closed prior to randomization
6. Patients with known metabolic bone disease (other than osteoporosis) which would negatively impact on the bone healing process.
7. Patients with known sensitivity to collagen.
8. Patients who are pregnant or breastfeeding at the time of study enrolment.
9. Patients currently being treated with radiation, chemotherapy, immunosuppression, or steroid therapy.
10. Patients receiving any other investigational drug or treatment.
11. Patients who have other injuries or conditions such as they are unable to communicate or consent

m)Patients with known breast or prostate cancer

f) Patients must be able and willing to provide informed consent, to complete study assessments, and to be followed for the period of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Estimated); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
cost analysis based on length of hospital stay, allograft, blood products and costs associated with complications and/ or re-admission. | 2 years

SECONDARY OUTCOMES:
Secondary efficacy end points will be the radiographic assessment of healing (RUST scale), the clinical assessment of weight-¬bearing status at 6 months post treatment, and the incidence of additional surgical/medical interventions to promote healing. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ross K Leighton, MD, Principal Investigator — CDHA
Locations (1):
- Halifax Infirmary, Halifax, Nova Scotia, Canada